CLINICAL TRIAL: NCT02846051
Title: Effect of Intensive Sports Practice on Lower Limb Varicose Veins
Acronym: VARISPORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Franche-Comté (Other)
Responsible Party: Principal Investigator, Laurent Mourot, MCU-HDR, University of Franche-Comté
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: EPSI_VARISPORT
Record Dates: First submitted 2016-07-15; First posted 2016-07-27 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Varicose Vein
Keywords: varicose vein; physical activity
MeSH Terms: conditions — Varicose Veins; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intensive sport practice (Other): intensive sport practice
  1. the subject must practice for more than six months a drive of at least 8 hours / week, intense, above the ventilatory threshold, or 60-70% of maximum consumption oxygen or 70-80% of maximum heart rate, ie beyond a moderate slowdown. If stopping the intensive sport practice, the duration of the stop at the time of the study should be less practice time.
  2. volunteers,
  3. from 18 to 80 years,
  4. free to consent.
  5. covered by social security.
  6. reported in the national register of healthy volunteers.
  The intervention is a lower limb venous examination = venous mapping
  Interventions: Procedure: venous mapping
- control group (Other): &) Volunteers who do not have intensive sport practice as it is defined in the group "intensive sport practice" 2) from 18 to 80 years, 3) free to consent. 4) covered by social security. 5) reported in the national register of healthy volunteers.
  The intervention is a lower limb venous examination = venous mapping
  Interventions: Procedure: venous mapping

INTERVENTIONS:
Procedure: venous mapping — clinical examination + doppler echo

SUMMARY:
Compare the frequency of varicose veins in the lower limbs in a population exposed to intensive sport compared to individuals matched by sex, age and body mass index (BMI) did not have an intensive sport.

DETAILED DESCRIPTION:
Chronic venous disease is a very common disease in industrialized countries. The prevalence of this disease is estimated in France 30.1% in men and 50.5% women.

Sufferers report pain, heaviness and itching of the lower limbs, and these symptoms are increased at night and in a warm environment. Clinically chronic venous disease resulting in varicose veins (veins visible under the skin, tortuous and dilated), edema (swelling predominant at the ankles) and in the later stages include skin damage of up 'to the ulcer.

The pathological mechanisms underlying chronic venous disease are mainly related to incontinence of the valves of the veins of the lower limbs. The initial role of these valves is to allow the return of blood to the heart and prevent it falls constantly in the legs. A breach of these valves therefore will result in an alteration of venous return and dilatation of the affected veins. It will be highlighted by a venous reflux when analyzing Doppler.

A number of parameters have been identified as factors favoring chronic venous disease in the lower limbs. Thus heredity (family history of venous disease), age, number of pregnancies among women, a history of phlebitis, overweight and physical inactivity increase the risk of chronic venous disease.

The effects of physical activity:

The practice of physical activity helps fight against physical inactivity. It is recognized as a protective factor against chronic venous disease. That is why the French and international companies of medicine and vascular surgery have incorporated in their recommendations to patients the practice of moderate physical activity and regular part of the prevention and treatment of chronic venous disease.

Moreover, the impact of intensive practice of a sport (versus "moderate and regular physical activity") of chronic venous disease is not known. Assumptions were issued from the nineteenth century on the possible risk of fostering the emergence of chronic venous disease at an excessive sports. Thus, from the 1820s Dr. Rima Thomas, surgeon of Napoleon's army, stated: "inertia as much as excessive activity come together to produce the same effect, the varicose vein." This idea is still relevant, in fact some experts recommend, at this time, intensive sports wear compression devices in the lower limbs during sports practice to prevent this phenomenon. However, no study has established a link between intensive practice of sport and venous condition of the legs.

The purpose of the study:

VARISPORT The study will aim to analyze the condition of the veins of the lower limbs in two groups of voluntary individuals, aged 18 to 80 years, in the same population:

* An "intensive sport practice": This group will consist of men and women who practice for more than 6 months, a drive of at least 8 hours / week, intense, above the ventilatory threshold, or 60-70 % maximum oxygen consumption or 70- 80% of maximum heart rate, ie beyond a moderate slowdown. If stopping the intensive sport practice, the duration of the stop at the time of the study should be less practice time.
* A "control" group: the subjects included in this group will have profiles that approximate subjects of the group "intensive practice sports", same sex, same age, BMI close; but the practice of a sport is less than 8 hours per week.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers
* From 18 to 80 years
* Free to consent
* Covered by social security
* Reported in the national register of healthy volunteers

Exclusion Criteria:

* Signed Refusal of the consent form .
* Refusal to be registered with the National File Healthy Volunteers.
* People exclusion period from another study
* Under guardianship
* Inability of the subject to hold long enough in standing position (20 minutes) for practicing phlebology examination.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2015-10; Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
varicose veins (C2 of the CEAP classification) | 3 years
  varicose vein definition : subcutaneous vein with a diameter greater than 3 mm while standing, usually winding, the seat of pathological reflux. Varicose veins may interest saphenous trunks, their tributaries and non saphenous network.
  Duplex Ultrasound Investigation of the Veins in Chronic Venous Disease of the Lower Limbs-UIP Consensus
  Chronic venous disorders Assessment Score (Carpentier PH, Poulain C, Fabry R, Chleir F, Guias B, Bettarel-Binon C. Ascribing leg symptoms to chronic venous disorders: the construction of a diagnostic score. J Vasc Surg Off Publ Soc Vasc Surg Int Soc Cardiovasc Surg North Am Chapter. nov 2007;46(5):991- 6.)

SECONDARY OUTCOMES:
lower limb vein calibers | 3 years
  echo doppler measurement of the antero posterior vein caliber
venous reflux | 3 years
  echo doppler Search venous reflux

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Tordi, PU, Study Director — Equipe d'Accueil 4267 : Fonctions et dysfonctions épithéliales Université de Franche Comté
Locations (1):
- Beliard, Besançon, France

IPD SHARING:
Plan to Share IPD: Yes
If a venous pathology is detected during this study, the data are passed on to the doctor of the subject